CLINICAL TRIAL: NCT00490412
Title: Randomized, Placebo-controlled Trial of the Safety and Effectiveness of Vitamin D Supplement to Improve Tubular Reabsorption of Phosphate and Decrease Bone Turnover in Adolescents and Young Adults With HIV Infection Being Treated With Antiretroviral Therapy Containing Tenofovir Compared to Those Being Treated With Antiretroviral Therapy Not Containing Tenofovir
Brief Title: Vitamin D Reabsorption in Adolescents and Young Adults With HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATN 063
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: Vitamin D; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: tenofovir/vitamin D (Experimental): Vitamin D3 (cholecalciferol), 50,000 IU as a single capsule, will be administered orally to subjects in Group A (who are already taking Tenofovir) once every four weeks during study visits.
  Interventions: Dietary Supplement: Vitamin D supplement
- B: tenofovir/placebo (Placebo Comparator): A placebo will be administered orally to subjects in Group B (who are already taking Tenofovir).
  Interventions: Other: Placebo
- C: no tenofovir/vitamin D (Experimental): Vitamin D3 (cholecalciferol), 50,000 IU as a single capsule, will be administered orally to subjects in Group C (who are not taking Tenofovir) once every four weeks during study visits.
  Interventions: Dietary Supplement: Vitamin D supplement
- D: no tenofovir/placebo (Placebo Comparator): A placebo will be administered orally to subjects in Group D (who are not taking Tenofovir).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D supplement — Vitamin D3 (cholecalciferol), 50,000 IU as a single capsule, will be administered orally to subjects in Groups A and C once every four weeks during study visits.
  Arms: A: tenofovir/vitamin D; C: no tenofovir/vitamin D
Other: Placebo — A placebo will be administered orally to subjects in Groups B and D once every four weeks during study visits.
  Arms: B: tenofovir/placebo; D: no tenofovir/placebo

SUMMARY:
The purpose of this study is to test the effects of Vitamin D on renal phosphate and bone loss, which are common in HIV infected adolescents and young adults being treated with tenofovir.

DETAILED DESCRIPTION:
ATN 063 tests the hypothesis that in a population of adolescents and young adults with HIV infection who are being treated with tenofovir as part of an antiretroviral (ARV) combination regimen, vitamin D supplementation will decrease renal phosphate loss, increase plasma phosphate, decrease plasma PTH, and improve markers of bone turnover, including a decrease in plasma N-telopeptide and BAP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and 0 days through 24 years and 364 days
* HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to study entry
* Currently being treated with a stable FDA-approved ARV combination therapy, containing > 3 antiretrovirals, for > 28 days, according to HRSA guidelines. Treatment regimen will not be started or changed for the purposes of participation in this study. Subjects will be receiving therapy at the direction of their treating physician
* Willingness to remain on the same ARV combination therapy for the 12-week duration of the study
* Ability and willingness to participate in the study by providing written informed consent
* Willingness to be randomized to receive either vitamin D or placebo

Exclusion Criteria:

* Prior hypersensitivity to vitamin D
* History of arteriosclerosis, renal stones, glomerulonephritis, nephrotic syndrome, or hypercalcemia
* Lactation or current pregnancy
* Active therapy for malignancy
* Known presence of gastrointestinal disease that would interfere with drug administration or absorption
* Serological evidence of Hepatitis B surface antigen (HBsAg)
* Confirmed creatinine clearance < 90 ml/min (calculated GFR from serum creatinine using the MDRD formula)
* Grade 3 or higher clinical toxicity

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To compare the change in renal tubular reabsorption of phosphate and markers of bone turnover. | Baseline, Week 4, Week 12
To measure the safety of 50,000 IU dose of vitamin D3 | Baseline, Week 4, and Week 8

SECONDARY OUTCOMES:
To measure the relationship of vitamin D plasma concentrations to renal tubular reabsorption of phosphate and markers of bone turnover | Baseline, Week 4, and Week 12
To measure the relationship of tenofovir exposure to renal tubular reabsorption of phosphate and markers of bone turnover | Baseline, Week 4, and Week 12
To measure the change in tenofovir exposure and creatinine clearance | Baseline, Week 4, and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Havens, M.S., M.D., Study Chair — Medical College of Wisconsin
Locations (15):
- United States (14):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical School, Baltimore, Maryland
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Havens PL, Hazra R, Stephensen CB, Kiser JJ, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 study team. Vitamin D3 supplementation increases fibroblast growth factor-23 in HIV-infected youths treated with tenofovir disoproxil fumarate. Antivir Ther. 2014;19(6):613-8. doi: 10.3851/IMP2755. Epub 2014 Feb 17. PMID 24535626
- [Derived] Havens PL, Kiser JJ, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Gordon CM, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 063 Study Team. Association of higher plasma vitamin D binding protein and lower free calcitriol levels with tenofovir disoproxil fumarate use and plasma and intracellular tenofovir pharmacokinetics: cause of a functional vitamin D deficiency? Antimicrob Agents Chemother. 2013 Nov;57(11):5619-28. doi: 10.1128/AAC.01096-13. Epub 2013 Sep 3. PMID 24002093
- [Derived] Havens PL, Stephensen CB, Hazra R, Flynn PM, Wilson CM, Rutledge B, Bethel J, Pan CG, Woodhouse LR, Van Loan MD, Liu N, Lujan-Zilbermann J, Baker A, Kapogiannis BG, Mulligan K; Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions 063 study team. Vitamin D3 decreases parathyroid hormone in HIV-infected youth being treated with tenofovir: a randomized, placebo-controlled trial. Clin Infect Dis. 2012 Apr;54(7):1013-25. doi: 10.1093/cid/cir968. Epub 2012 Jan 19. PMID 22267714
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org